CLINICAL TRIAL: NCT03998189
Title: Pilot Study: Metabolic and Microbial Profiling of Lung Cancer
Brief Title: Metabolic and Microbial Profiling of Lung Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study deemed no longer feasible
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00059167; WFBCCC 03219 (Other: Wake Forest Baptist Comprehensive Cancer Center); P30CA012197 (NIH)
Record Dates: First submitted 2019-06-20; First posted 2019-06-26 (Actual); Results first posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Nonsmall Cell Lung Cancer; Nonsmall Cell Lung Cancer Stage
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Blood Specimen Collection; Urine Specimen Collection

STUDY DESIGN:
Intervention Model Description: 45 female/ 45 male participants
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Female Participants (Experimental): 45 female patients will be screened to participate.
  Interventions: Other: Breath Collection; Other: Saliva Collection; Other: Blood Collection; Other: Urine Collection; Other: Tumor Collection; Other: Medical History Data Collection
- Male Participants (Experimental): 45 male patients will be screened to participate
  Interventions: Other: Breath Collection; Other: Saliva Collection; Other: Blood Collection; Other: Urine Collection; Other: Tumor Collection; Other: Medical History Data Collection

INTERVENTIONS:
Other: Breath Collection — Pre-surgery, two 500 ml of exhaled breath volatiles (EBV) in each of 4 collection tubes will be collected in 5-7 min of breathing
Other: Saliva Collection — Pre-surgery, 2 ml minimum of saliva will be collected into SalivaBio Passive Drool collection tubes
Other: Blood Collection — Pre-surgery, an optional 5 ml blood sample in each redtop and purple top vacutainer blood collection tube
Other: Urine Collection — Pre-surgery, 25 ml minimum of urine will be collected in sterile specimen containers
Other: Tumor Collection — During surgical tumor removal, a tumor tissue sample will be collected
Other: Medical History Data Collection — Medical history will be obtained from the patients charts to identify demographics (age, race, ethnicity, zip code), oncologic history (date of diagnosis and cancer type), and medical history of disease.

SUMMARY:
This pilot study will establish non-invasive sample collections, including breath, saliva, blood and urine pre-surgery and at the participant's one-month post-surgery follow-up visit. Participants with suspected non-small cell lung cancer (NSCLC) stage I-III will be recruited.

DETAILED DESCRIPTION:
Primary Objective

* To evaluate the feasibility of adding non-invasive sample collections in the pre-surgical setting and at the post-surgery follow-up visit.
* To identify and assess metabolic and microbial signatures collected at pre- and post-surgery and determine which are indicative of lung cancer.

Secondary Objective

* To identify signatures which are associated with lung cancer stage.
* To identify signatures which are impacted by patient's pulmonary function status.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients age >18 years, of all racial and ethnic origins, with suspected nonsmall cell lung cancer stages I, II, and III, as evident through radiographic evidence and felt acceptable to undergo surgical resection.
* Patients who have the ability to understand and the willingness to sign a written consent form.

Exclusion Criteria:

* Patients who are have taken antibiotics within two weeks.
* Patients who are on continuous supplemental oxygen.
* Patients currently undergoing active treatment for other malignancies.
* Subjects who are unable or unwilling to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Bishop, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Female Participants | Male Participants
Started | 0 | 1
Completed | 0 | 0 (Samples were collected but were not analyzed as the analysis would have been done once a proper batch of samples were collected. This did not occur as the study was found to no longer be feasible and was terminated.)
Not Completed | 0 | 1
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Population: There were no female participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Female Participants | Male Participants | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Customized [Number; unit: years]
  Enrolled participant |  | 82 | 82
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 0 | 0
  Male |  | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 | 0
  Not Hispanic or Latino |  | 1 | 1
  Unknown or Not Reported |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 0 | 0
  White |  | 1 | 1
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Needed for Feasibility
Description: The primary objectives is to assess the feasibility of adding these non-invasive sample collections to pre- and post-surgery visits the following outcomes (counts) will be gathered - (number eligible for trial, number that consent to participate, number that provide pre-surgery samples, number that provide post-surgery samples) using a 95% exact Clopper-Pearson confidence interval for each feasibility estimate.
Time Frame: One month
Population: Biosamples that were collected were not analyzed as the analysis would be done once a proper batch of samples were collected. Given that never happened, investigators have no study results to report.
Arm/Group | Female Participants | Male Participants
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Pre-Surgery and Post-Surgery Metabolic Signatures
Description: Metabolic assessments will be taken before and after surgery of lung cancer biomarkers to examine a series of paired t-tests to determine which markers significantly change between the two time points for participants.
Time Frame: One month post surgery
Population: as for outcome 1
Arm/Group | Female Participants | Male Participants
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Pre-Surgery and Post-Surgery Microbial Signatures
Description: as for outcome 2
Time Frame: One month post surgery
Population: as for outcome 1
Arm/Group | Female Participants | Male Participants
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Identification of Lung Cancer Stage Specific Signatures
Description: For lung cancer examine whether pre-surgery, post-surgery or change from pre- to post- surgery metabolic or microbial measures are different depending on lung cancer stage. Consideration of the metabolic or microbial measures as outcomes and use a general linear models framework to see if lung cancer stage (included as a class variable, but then examined as an ordinal variable using a contrast statement in general linear model) is associated with any marker.
Time Frame: One month post surgery
Population: as for outcome 1
Arm/Group | Female Participants | Male Participants
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Identification of Signatures Associated With Pulmonary Function
Description: For pulmonary function, the same approach as for lung cancer stage, except that pulmonary function will be considered as a continuous variable in the model. Pulmonary function can be examined at both time-points (pre- and post- surgery) thus we can examine the relationships between pulmonary function measures and biomarker measures at each time points (and the change in measures over time).
Time Frame: One month post surgery
Population: as for outcome 1
Arm/Group | Female Participants | Male Participants
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: There were no female participants enrolled on this study before it was terminated.
Arm/Group | Female Participants | Male Participants
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-03): https://cdn.clinicaltrials.gov/large-docs/89/NCT03998189/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/89/NCT03998189/ICF_001.pdf